CLINICAL TRIAL: NCT05445414
Title: A Mobile App Serious Game to Increase Public Awareness of Appropriate Antibiotic Use in the Community
Brief Title: A Mobile App Serious Game to Increase Awareness of Antibiotic Use in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: National Healthcare Group Polyclinics (Other Government); Temasek Polytechnic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FY2022HZ
Record Dates: First submitted 2022-06-27; First posted 2022-07-06 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Antimicrobial Resistance

STUDY DESIGN:
Intervention Model Description: A two-arm randomised controlled trial with the intervention group receiving an educational app and the control group not receiving any app intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants randomized to the intervention group will be asked to use the "SteWARdS Antibiotic Defense" app-an evidence-based serious game app developed by the study team-for a minimum of five days. They will also need to complete three sets of questionnaires - one set at baseline, one set after completing the quest in the app, and another set 6-10 weeks after they complete the quest in the app.
  Interventions: Device: "SteWARdS Antibiotic Defense" app
- Control group (No Intervention): Participants randomized to the intervention group would be asked to complete two sets of questionnaires - one set at baseline and another set 6-10 weeks later.

INTERVENTIONS:
Device: "SteWARdS Antibiotic Defense" app — The "SteWARdS Antibiotic Defense" app is an evidence-based serious game app developed by the study team. The app uses gamification theories to increase user engagement and to deliver bite-sized information to participants. For example, players will learn about the uses of antibiotics through the messages delivered through the game and the cost of tackling antibiotic-resistant infections through purchasing an expensive antibiotic with the virtual currency earned from the games.
  Arms: Intervention group

SUMMARY:
The widespread and unnecessary use of antibiotics has encouraged the growth of antibiotic-resistant bacteria which can cause hard-to-treat and deadly infections. These infections are due to antimicrobial resistance (AMR). The public's lack of knowledge on the indication for and proper use of antibiotics often leads to unnecessary patient demands and subsequent misuse of antibiotics. Traditional mass public educational efforts through the use of brochures, posters and advertisements are extensive in outreach but questionable in effectiveness in improving the general public's knowledge on appropriate antibiotics use and AMR.

Serious games app provides an additional venue for public education outreach to the population since a substantial amount of time is spent using smartphones. The use of serious games is expected to increase user engagement in learning, which will lead to short- and long-term improvements in knowledge, attitudes and perceptions on the appropriate use of antibiotics.

The study team has co-developed an evidence-based serious game app- "SteWARdS Antibiotic Defense" -with Temasek Polytechnic. Users will be brought on a quest to learn about antibiotic use and AMR through mini-games and the bite-sized information released throughout the game quest. We intend to clinically validate our evidence-based app and improve its application with actual participants' feedback on its usage. Hence, this study aims to evaluate the effectiveness of an evidence-based serious game mobile application (SteWARdS Antibiotic Defense) in improving the knowledge on, attitude towards, and perception (KAP) of appropriate antibiotic use and AMR among Singaporeans.

The primary objective is to assess the change in knowledge on antibiotic use and AMR among the app users compared with the control group. The secondary objectives are to:1) Assess the extent of user engagement of the app by evaluating the users' average screen time per day; and 2) Assess the level of user satisfaction in using the app for learning through a user satisfaction survey.

DETAILED DESCRIPTION:
The widespread and unnecessary use of antibiotics has accelerated the development of antimicrobial resistance (AMR) which can cause infections that are fatal and resistant to treatment. One pertinent factor contributing to the misuse of antibiotics is the public's knowledge deficit of the indication for and proper use of antibiotics. This knowledge deficit often leads to unnecessary patient demand for antibiotics and subsequent misuse of them. The public has low awareness of the gravity of AMR as it appears to be a non-imminent life-threatening problem. Traditional mass public educational efforts through the use of brochures, posters and advertisements are extensive in outreach but questionable in effectiveness in improving the general public's knowledge on appropriate antibiotics use and AMR.

Serious games app provides an additional venue for public education outreach to the population since a substantial amount of time is spent using smartphones. Leveraging digital technology to increase the awareness of antimicrobial resistance and the knowledge of appropriate antibiotic use is timely as Singapore develops into a smart nation. The use of serious games is postulated to increase user engagement in learning, which will lead to short- and long-term improvements in knowledge, attitudes and perceptions on the appropriate use of antibiotics.

The study team has co-developed an evidence-based serious game app- "SteWARdS Antibiotic Defense" -with Temasek Polytechnic. Users will be brought on a quest to learn about antibiotic use and AMR through mini-games and the bite-sized information released throughout the game quest. We intend to clinically validate our evidence-based app and improve its application with actual participants' feedback on its usage. Hence, this study aims to evaluate the effectiveness of an evidence-based serious game mobile application (SteWARdS Antibiotic Defense) in improving the knowledge on, attitude towards, and perception (KAP) of appropriate antibiotic use and AMR among Singaporeans.

The primary objective is to assess the change in knowledge on antibiotic use and AMR among the app users compared with the control group. The secondary objectives are to:1) Assess the extent of user engagement of the app by evaluating the users' average screen time per day; and 2) Assess the level of user satisfaction in using the app for learning through a user satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 65 years
* Have access to an Android smartphone
* Able to comprehend the English language

Exclusion Criteria:

* Unable to install Android mobile applications
* Not proficient with using smartphone applications
* Cognitive or visual impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in the knowledge, attitudes, and perception of participants towards antibiotics use. | Baseline, immediate completion of intervention, 6-10 weeks post intervention
  Change in the knowledge, attitudes, and perception of participants towards antibiotics use and AMR at 6-10-weeks post-intervention from the baseline, measured by the survey. The immediate knowledge change will be measured by the in-app questionnaire knowledge questions, post-completion of the game quest.

SECONDARY OUTCOMES:
User engagement level | Five days - 2 weeks
  The time spent on the app each day, tracked by the study team backend
Satisfaction level of playing the games in the app | Immediately completing the game quest in the app
  Satisfaction level of playing the games in the app after completing the game quest via a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Zhilian Huang, Ph.D, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Ang Mo Kio Polyclinic, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers to ensure participants' data confidentiality.

REFERENCES:
- [Derived] Huang Z, Ow JT, Tang WE, Chow A. An Evidence-Based Serious Game App for Public Education on Antibiotic Use and Resistance: Randomized Controlled Trial. JMIR Serious Games. 2024 Sep 5;12:e59848. doi: 10.2196/59848. PMID 39235853
- [Derived] Huang Z, Tang WE, Guo H, Natarajan K, Lee TH, Yeo TW, Chow A. An Evidence-Based Serious Game App for Public Education on Antibiotic Use and Antimicrobial Resistance: Protocol of a Randomized Controlled Trial. JMIR Res Protoc. 2023 Mar 28;12:e45833. doi: 10.2196/45833. PMID 36976619